CLINICAL TRIAL: NCT01076569
Title: Target: Identification for High Risk Childhood AML Based on Genome-Wide Analysis
Brief Title: Biomarkers in Bone Marrow Samples From Pediatric Patients With High-Risk Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B14; NCI-2011-02212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AAML10B14 (Other: Children's Oncology Group); AAML10B14 (Other: Children's Oncology Group); AAML10B14 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Acute Basophilic Leukemia; Childhood Acute Eosinophilic Leukemia; Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Minimally Differentiated Myeloid Leukemia (M0); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Recurrent Childhood Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Eosinophilic, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (molecular analysis): Banked bone marrow samples from diagnosis and remission are used to develop a detailed molecular map of pediatric high-risk acute myeloid leukemia. Analysis includes genome SNP genotyping, expression, and methylation profiling.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot research trial studies biomarkers in bone marrow samples from pediatric patients with high risk acute myeloid leukemia. Studying samples of bone marrow from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide a detailed, molecular map of pediatric high risk acute myeloid leukemia (AML).

II. To identify mutations, expression profile, gene copy number, loss of heterozygosity (LOH) status and genomic methylation patterns in order to identify novel changes associated with pediatric AML.

III. To generate fibroblast cell lines in order to obtain germline nucleic acids from marrow specimens from AML patients with induction failure.

IV. To identify genomic alterations contributing to induction failure in childhood AML.

OUTLINE:

Banked bone marrow samples from diagnosis and remission are used to develop a detailed molecular map of pediatric high-risk acute myeloid leukemia. Analysis includes genome single nucleotide polymorphism (SNP) genotyping, expression, and methylation profiling.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia

  * High-risk disease
* Treated on COG-AAML03P1 or COG-AAML0531
* Meets the following criteria:

  * Initial remission with no known adverse risk factors
  * High quantity and quality of ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) available
  * Highly enriched specimens with >= 50% blast available

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any patient with a diagnosis of acute myeloid leukemia meeting the other criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Detailed molecular map of pediatric high-risk acute myeloid leukemia | Baseline
Mutations in identifying novel changes associated with pediatric AML | Baseline
Expression profile in identifying novel changes associated with pediatric AML | Baseline
Gene copy number in identifying novel changes associated with pediatric AML | Baseline
LOH status in identifying novel changes associated with pediatric AML | Baseline
Genomic methylation patterns in identifying novel changes associated with pediatric AML | Baseline
Genomic and transcriptome alterations associated with induction failure | Baseline
Genomic alterations contributing to induction failure in childhood AML | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Meshinchi, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States